CLINICAL TRIAL: NCT03033849
Title: User Performance Evaluation of Contour® Next One, Accu-Chek® Aviva Connect, FreeStyle Freedom Lite, OneTouch® Verio and GlucoMen® Areo Blood Glucose Monitoring Systems Following ISO 15197:2013
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut für Diabetes-Technologie Forschungs- und Entwicklungsgesellschaft mbH an der Universität Ulm (Other)
Collaborators: Ascensia Diabetes Care (Industry)
Responsible Party: Sponsor
Other Study IDs: IDT-1608-AL
Record Dates: First submitted 2017-01-16; First posted 2017-01-27 (Estimated); Last update posted 2017-09-12 (Actual); Status verified 2017-09

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

ARMS (1):
- Blood glucose measurement (Experimental): Every study subject shall test three out of the five devices. The testing order of the BGMS will be changed on each subject to minimize any order effects on measurement results.
  Interventions: Device: Blood glucose monitoring system for self-testing Contour® Next One; Device: Blood glucose monitoring system for self-testing Accu-Chek® Aviva Connect; Device: Blood glucose monitoring system for self-testing FreeStyle Freedom Lite; Device: Blood glucose monitoring system for self-testing OneTouch® Verio; Device: Blood glucose monitoring system for self-testing GlucoMen® areo

INTERVENTIONS:
Device: Blood glucose monitoring system for self-testing Contour® Next One — This is a user performance study, that is intended to show whether people with diabetes are able to obtain accurate measurement results with a blood glucose monitoring system (BGMS).
  The subjects' measurement technique (e.g. applying blood onto the system reagent, reading the result) will be observed and documented by study personnel.
  Immediately after the measurement by the subject, the study personnel will perform a measurement with the same test meter.
  Measurement results obtained by the subjects with the BGMS will be compared to measurement results obtained with the comparison method.
  Sample collection for the comparison measurement will be performed by study personnel within 5 min after the subject's measurement with the test meter.
  The samples will be collected from the subjects' skin puncture (if possible), an additional skin puncture (if required) will be documented.
  An additional skin puncture will be performed by study personnel with single-use lancing devices.
  Other Names: Contour® Next One, Accu-Chek® Aviva Connect, FreeStyle Freedom Lite, OneTouch® Verio, GlucoMen® areo
Device: Blood glucose monitoring system for self-testing Accu-Chek® Aviva Connect
Device: Blood glucose monitoring system for self-testing FreeStyle Freedom Lite
Device: Blood glucose monitoring system for self-testing OneTouch® Verio
Device: Blood glucose monitoring system for self-testing GlucoMen® areo

SUMMARY:
The user performance evaluation shows whether people with diabetes are able to obtain accurate measurement results with a blood glucose monitoring system. In this study, user performance evaluation will be performed for Contour® Next One (Ascensia Diabetes Care GmbH), Accu-Chek® Aviva Connect (Roche Diabetes Care GmbH), FreeStyle Freedom Lite (Abbott Diabetes Care Inc.), OneTouch® Verio (LifeScan Europe) and GlucoMen® areo A. Menarini Diagnostics S.r.l. (based on ISO 15197:2013; EN ISO 15197:2015, clause 8.

For each BGMS, measurement procedures for user performance evaluation will be performed with 1 test meter and 1 reagent system lot by the study subjects.

The same meter and an additional test meter will be used for double measurements performed by study personnel (with the same reagent system lot used by subjects).

ELIGIBILITY:
Inclusion Criteria:

* Male or female, with type 1 diabetes, type 2 diabetes or subjects without diabetes
* Signed informed consent form
* Minimum age of 18 years
* Subjects are legally competent and capable to understand character, meaning and consequences of the study.
* If blood glucose values < 80 mg/dl or > 300 mg/dl shall be measured after short term alteration in insulin therapy:
* Male or female with type 1 diabetes and intensified insulin therapy or insulin pump therapy.
* Signature of subjects to document consent with these procedures on informed consent form.

Exclusion Criteria:

* Pregnancy or lactation period
* Severe acute disease (at the study physician's discretion)
* Severe chronic disease with potential risk during the test procedures (at the study physician's discretion)
* Current constitution that compromises the subject's capability to participate in the study (at the study physician's discretion)
* Being unable to give informed consent
* < 18 years
* Legally incompetent
* Being committed to an institution (e.g. psychiatric clinic)
* Language barriers potentially compromising an adequate compliance with study procedures
* Dependent on investigator or sponsor
* If blood glucose values < 80 mg/dl shall be measured after short term alteration in insulin therapy, subjects with type 1 diabetes, suffering from:
* Coronary heart disease
* Condition after myocardial infarction
* Condition after cerebral events
* Peripheral arterial occlusive disease
* Hypoglycemia unawareness

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2017-01; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Acceptance criteria defined by ISO 15197:2013 (E) will be applied | For each subject, the experimental phase has an expected duration of up to 3 hours
  95 % of the individual glucose measured values shall fall within ± 15 mg/dl (0.83 mmol/l) of the measured values of the comparison measurement procedure at glucose concentrations < 100 mg/dl (5.55 mmol/l) and within ± 15 % at glucose concentrations ≥ 100 mg/dl (5.55 mmol/l).

CONTACTS AND LOCATIONS:
Locations (1):
- Institut für Diabetes-Technologie Forschungs- und Entwicklungsgesellschaft mbH an der Universität Ulm, Ulm, Baden-Wurttemberg, Germany

REFERENCES:
- [Derived] Jendrike N, Baumstark A, Pleus S, Liebing C, Kamecke U, Haug C, Freckmann G. Accuracy of five systems for self-monitoring of blood glucose in the hands of adult lay-users and professionals applying ISO 15197:2013 accuracy criteria and potential insulin dosing errors. Curr Med Res Opin. 2019 Feb;35(2):301-311. doi: 10.1080/03007995.2018.1491832. Epub 2018 Jul 19. PMID 29927663